CLINICAL TRIAL: NCT05650892
Title: Male-female Differences in Immunohistological and Biomechanical Properties of the Thoracic Aorta
Acronym: MAFATS
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hanneke Takkenberg (Other)
Responsible Party: Sponsor-Investigator, Hanneke Takkenberg, Prof. dr., Erasmus Medical Center
Organization: Erasmus Medical Center (Other)
Other Study IDs: MEC-2020-0085
Record Dates: First submitted 2022-06-07; First posted 2022-12-14 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2023-02

CONDITIONS: Thoracic Aortic Aneurysm
MeSH Terms: conditions — Aortic Aneurysm, Thoracic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Thoracic aorta (residual tissue).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Sample collection aortic tissue: Sample collection thoracic aorta tissue

SUMMARY:
Thoracic aortic aneurysms (TAA) result from progressive dilatation of the thoracic aorta and confer a risk for aortic dissection or rupture, which is associated with significant morbidity and mortality. In the Netherlands there are an estimated 200.000 adults with TAA, and annually 600 deaths after aortic dissection or rupture. There are clear differences in the incidence of TAA between men and women, with a higher incidence in men. Little is known on possible differences in outcome between male and female patients with Thoracic Aortic Aneurysm (TAA). Aortic disease is thought to affect men more frequently than women, and aortic growth is different between men and women. Current data suggest that women are at an increased risk of both dying from aortic dissection and having aorta-related complications compared to men (1). The mechanisms for these male-female difference in TAA outcome remain, however, unclear. The timing of preventive surgery is now not different for men and women, but gender-based cut-off values for maximal aortic diameter based on differences in vessel wall composition might be needed.

DETAILED DESCRIPTION:
Thoracic aortic aneurysms (TAA) result from progressive dilatation of the thoracic aorta and confer a risk for aortic dissection or rupture, which is associated with significant morbidity and mortality. In the Netherlands there are an estimated 200.000 adults with TAA, and annually 600 deaths after aortic dissection or rupture. There are clear differences in the incidence of TAA between men and women, with a higher incidence in men. Little is known on possible differences in outcome between male and female patients with Thoracic Aortic Aneurysm (TAA). Aortic disease is thought to affect men more frequently than women, and aortic growth is different between men and women. Current data suggest that women are at an increased risk of both dying from aortic dissection and having aorta-related complications compared to men(1). However, the mechanisms for these male-female differences in TAA outcome remain unclear. The timing of preventive surgery is not different for men and women, but gender-based cut-off values for maximal aortic diameter based on differences in vessel wall composition might be beneficial for outcome.

The current research project aims to implement male-female specific insights into aortic root and ascending aorta characteristics into clinical practice, allowing better identification of high risk Thoracic Aortic Aneurysm (TAA) patients and better timing of intervention. With this study the investigators aim to obtain insight into male-female differences in the immunohistological and biomechanical properties of the thoracic aortic wall. In order to reveal possible mechanisms for male-female differences in TAA.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥ 18 years old) who have a thoracic aortic aneurysm and are scheduled for elective thoracic aortic surgery in the Erasmus MC or the LUMC.

Exclusion Criteria:

* Patients with a known connective tissue disease (e.g. Marfan Syndrome and Ehlers-Danlos syndromes).
* Connective tissue disease,

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults (≥18 years old) who will undergo or already underwent elective surgery for thoracic aortic aneurysm at Erasmus MC, Rotterdam and LUMC, Leiden.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-12-16 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Male-female differences in immunohistochemical and mass spectrometry-based estrogen and testosterone receptor expression levels (and density) in the proximal aortic wall | 1 year
  To investigate male-female differences in estrogen receptor (ESR-alpha and ESRbeta) and testosterone receptor (AR) tissue expression in the wall of the aortic root and ascending aorta by immunohistochemical techniques and mass spectometry. Comparisons will be made using a students t-test.

SECONDARY OUTCOMES:
Male-female differences in immunohistochemical or mass spectrometry-based sex hormone receptor expression levels (and density) in the proximal aortic wall. | 1 year
  To perform an explorative analysis of differences in sex hormone receptor expression in the relation to 1) the immunohistological properties of the aortic wall structure (smooth muscle cell differentiation, presence of macrophages, endothelial cell activation and extracellular matrix, through the following markers: alpha smooth muscle actin, sex hormone receptors (ESR1, RAGE, MMP 2, 3 and 9 and aromatase expression as marker for estrogen synthesis in SMC in both male and female), presence of macrophages (CD68 and MAC2) and endothelial cell activation (NOS3, TGF-β signaling) and extracellular matrix (a.o. fibrillin 1, elastin, collagen and crosslinking)) and to (1) sex hormone (androstenedione, DHEA, testosterone and SHBG in nmol/L, LH and FSH in IU/L, DHEA-S in micromole/L, AMH in micrograms/L, estradiol in picomol/L) and sRAGE (picograms/L) levels in blood, (2) aortic diameter (in millimeters) and (3) age (in years) using linear regression models.

CONTACTS AND LOCATIONS:
Overall Officials: Hanneke Takkenberg, Prof. dr., Principal Investigator — Erasmus Medical Center
Locations (1):
- Erasmus MC, Rotterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
All our anonymised individual patient data (IPD) will be available to other researchers, upon reasonable request and after publication of the manuscript. This includes IPD derived from all analyses that were performed for and used in this study.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will become available upon request after a period of twelve months from the date of publication. The length of availability of IPD will depend on and therefore be based on the request of the researchers.
Access Criteria: IPD will be shared with scientific researchers and is dependent on the research questions. The analysis and interpretation by the researcher will be checked by the project leader before any submission of the manuscript.